CLINICAL TRIAL: NCT01803971
Title: Obtaining Vascular Access (Venous or Intraosseous) During Cardiac Arrest in Out-of-hospital Care: Delays and Failure Risk Factors
Brief Title: Cardiac Arrest and Intra Osseous Infusion
Acronym: ACCIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2011/13; 2010/080 (Other: USMR / Edelweiss)
Record Dates: First submitted 2013-01-16; First posted 2013-03-04 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; peripheral venous access; intraosseous access
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vascular access in out-of-hospital cardiac arrest patients (Experimental): Obtention of vascular access according to the current strategy, ie after one unsuccessful attempt to obtain a peripheral venous access, use of an intra osseous device
  Interventions: Other: Obtention of vascular access in out-of-hospital cardiac arrest patients according to the current strategy

INTERVENTIONS:
Other: Obtention of vascular access in out-of-hospital cardiac arrest patients according to the current strategy — Current strategy of obtention of a vascular access : first attempt by peripheral venous access and if failure switch to intraosseous route

SUMMARY:
the international recommendations don't explain the place of the intraosseous infusion in the reanimation of adult cardiac arrest; the goal of this preliminary study is to inform the delay for obtaining a vascular access by evaluation of a current strategy (using intraosseous infusion after one peripheral venous access failure) and to determine the potential failure risk factors of venous access.

DETAILED DESCRIPTION:
In 2010, the European Resuscitation Council and the International Liaison Commitee on Resuscitation have made new recommendations about management of cardiac arrest. The intraosseous infusion was described as an alternative to the peripheral venous access, before the intra tracheal way for adrenaline administration. But this work doesn't specify the delay and the circumstance for this use: time to obtain a vascular access, number of failure, difficulty to obtain a venous access. Furthermore the recent improvements in intraosseous devices may make it relevant to compare intra osseous infusion and venous access in first intention in adult's cardiac arrest in view of the significant number of venous failures and of the subsequent delay of adrenaline administration.

The goal of this preliminary study is to inform the delay to obtain a vascular access by evaluation of a current care (using intravenous infusion after one peripheral venous access failure) and to determine the potential failure's risk factors of venous access.

Main objective: estimate the delay to obtain an effective vascular access (peripheral venous access, intra osseous infusion, central venous access) in resuscitation of adult's cardiac arrest by out of hospital care unit according to the international recommendations.

Study design: monocentric prospective cohort of consecutive patients presenting with out-of-hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or over
* patients insured by social security
* cardiac arrest (all causes) with mobilisation of a intensive mobile care unit in primary intervention
* medical resuscitation indicated

Exclusion Criteria:

* pregnancy
* contraindication osseous infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
functional vascular access | at inclusion (day 0)
  time for obtaining a functional vascular access from the beginning of out-of-hospital cardiac arrest management

CONTACTS AND LOCATIONS:
Overall Officials: Paul PEREZ, MD, PhD, Study Chair — University Hospital Bordeaux, France; Bruno SIMONNET, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- CHU Bordeaux, Bordeaux, France